CLINICAL TRIAL: NCT04181242
Title: Epidemiology of Injuries in Elite Badminton Players: a Prospective Study
Acronym: BADINSEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: BADINSEP
Record Dates: First submitted 2019-11-23; First posted 2019-11-29 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2019-11

CONDITIONS: Sport Injury
Keywords: Epidemiology, Incidence, Athletic Injuries, Racquet Sports, Badminton
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: To determine the incidence and characteristics of injuries in elite badminton players over a competitive season.

Design: 12-months prospective cohort study Setting: The French National Institute of Sport, Expertise, and Performance (INSEP).

Participants: Twenty international elite badminton players Independent variables: The type, the location, the occurrence of the injury (match or training), the footwork type, the type of shot and the perceived fatigue were collected.

Main Outcome Measures: Injury incidence rates were calculated per 1000 hours of play (Hop).

ELIGIBILITY:
Inclusion Criteria:

* Badminton players training at the at the French National Institute of Sport, Expertise, and Performance (INSEP)
* Participant competing at an international level
* Medical follow-up over the 12-months duration of the study

Exclusion Criteria:

* Participant unable to speak and read French language
* Participant under the age of 18
* Lack of informed and signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the international elite badminton players training at the at the French National Institute of Sport, Expertise, and Performance (INSEP)
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Injury incidence rates | Injury incidence rates were calculated per 1000 hours of play (Hop) over the 12-month prospective follow-up
  Injury incidence rates were calculated per 1000 hours of play (Hop).

SECONDARY OUTCOMES:
Injury incidence rates according to gender | Injury incidence rates were calculated per 1000 hours of play (Hop) over the 12-month prospective follow-up
  Injury incidence rates were calculated per 1000 hours of play (Hop) in male and female
Injury incidence rates according to discipline | Injury incidence rates were calculated per 1000 hours of play (Hop) over the 12-month prospective follow-up
  Injury incidence rates were calculated per 1000 hours of play (Hop) in singles and doubles players
Injury incidence rates according to occurence | Injury incidence rates were calculated per 1000 hours of play (Hop) over the 12-month prospective follow-up
  Injury incidence rates were calculated per 1000 hours of play (Hop) in match or training
Description of injuries according to location (on the body, n) | Description of the number of injuries according to location of the injury on the body (n) over the 12-month prospective follow-up
  Number of injuries according to location of the injury (on the body, n)
Description of injuries according to type of the injury (n) | Description of injuries according to the type of the injury (structure: muscle, tendon, bone, nerve...) (n) over the 12-month prospective follow-up
  Number of injuries according to type of the injury (n)
Description of injuries according to location (on the body, % of all) | Description of the distribution of injuries according to location of the injury on the body (%) over the 12-month prospective follow-up
  Distribution of injuries according to location of the injury (on the body, % of all)
Description of injuries according to type of the injury (% of all) | Description of the distribution of injuries according to the type of the injury (structure: muscle, tendon, bone, nerve...) (%) over the 12-month prospective follow-up
  Distribution of injuries according to type of the injury (% of all)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided